CLINICAL TRIAL: NCT02423187
Title: Rabeprazole Specific Clinical Experience Investigation for the Long-term Combination Therapy With Low-dose Aspirin
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: PRT12T
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Gastric Ulcer; Duodenal Ulcer
Keywords: Stomach ulcer; Duodenal ulcer; Rabeprazole; Recurrence
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Arm 1: Participants with combination therapy (rabeprazole and low-dose aspirin)
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention

SUMMARY:
To investigate the safety and efficacy of long-term combination therapy with rabeprazole and low-dose aspirin.

ELIGIBILITY:
Inclusion criteria:

1. Patients taking long-term low-dose aspirin for prevention of thrombus/embolism at the start of administration of rabeprazole (including patients who start low-dose aspirin on the same day as the start of administration of rabeprazole).
2. Patients with a history of gastric/duodenal ulcers.
3. Patients requiring long-term use of rabeprazole for prevention of recurrence of gastric/duodenal ulcers induced by low-dose aspirin.

Exclusion criteria:

1. Patients with gastric/duodenal ulcers at the start of administration of rabeprazole.
2. Patients with active upper gastrointestinal bleeding at the start of administration of rabeprazole.
3. Patients with contraindication for rabeprazole.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with long-term combination therapy with low-dose aspirin
Sampling Method: Non-Probability Sample
Enrollment: 1568 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions | 52 weeks

SECONDARY OUTCOMES:
Recurrence rate of peptic ulcer | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katsuya Sugizaki, Study Director — Drug Fostering and Evolution Coordination Department, Corporate Medical Affairs Headquarters, Eisai Co., Ltd.
Locations (3):
- Japan (3):
  - Nagoya
  - Osaka
  - Tokyo